CLINICAL TRIAL: NCT01224717
Title: A Phase I, Partially Blinded, Randomized, Placebo Controlled, Active Comparator Study to Explore the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics in Post-menopausal Women After Daily Oral Doses of PTH134
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral Doses of PTH134 in Post-menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharamceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPTH134A2102; 2009-015933-64 (EudraCT Number)
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Post-menopausal Osteoporosis
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- PTH134 (Experimental)
  Interventions: Drug: PTH134
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Forsteo (Active Comparator)
  Interventions: Drug: Forsteo

INTERVENTIONS:
Drug: PTH134
  Arms: PTH134
Drug: Placebo
  Arms: Placebo
Drug: Forsteo
  Arms: Forsteo

SUMMARY:
This study is designed to provide information about the bone-anabolic response of PTH134 when administered orally, in comparison to Forsteo®, the sub-cutaneous form of teriparatide, the active ingredient in PTH134.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women osteoporotic/osteopenic with an additional risk factor 45 to 80 years old

Exclusion Criteria:

* Use of estrogen or hormone replacement therapy
* Use of parathormone or parathormone fragments, calcitonin, aluminum supplements, within 12 months prior to first dose.
* Use of bisphosphonates and strontium ranelate
* Cancer or history of malignancy of any organ system
* Any radiation therapy to the skeleton.
* Any known clinically significant disease affecting calcium metabolism. Any history of metabolic disorders including Paget's disease, osteogenesis imperfecta, or osteomalacia.
* History or clinical evidence of any impairment of thyroid function
* Other protocol-defined inclusion/exclusion criteria apply.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measure: Effects of treatment on bone biomarkers. Measure levels of PINP, CTX-1, and serum calcium levels, serum phosphate, P1CP, bone-specific alkaline phosphatase, osteocalcin. | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in serum calcium levels after 12 weeks of treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Denmark (2):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Ballerup Municipality
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Munich